CLINICAL TRIAL: NCT00830960
Title: A Comparison of Platelet Inhibition Following Prasugrel or Clopidogrel Administration in Asian Acute Coronary Syndrome Subjects Who Are to Undergo Percutaneous Coronary Intervention
Brief Title: A Comparison of Antiplatelet Therapies in Asian Subjects With Acute Coronary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11299; H7T-MC-TACE (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Results first posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Prasugrel 60/10 Primary (Experimental): Loading dose 60 mg followed by maintenance dose 10 mg/day
  Interventions: Drug: Prasugrel
- Prasugrel 30/7.5 Primary (Experimental): Loading dose 30 mg followed by maintenance dose 7.5 mg/day
  Interventions: Drug: Prasugrel
- Prasugrel 30/5 Primary (Experimental): Loading dose 30 mg followed by maintenance dose 5 mg/day
  Interventions: Drug: Prasugrel
- Clopidogrel 300/75 Primary (Active Comparator): Loading dose 300 mg followed by maintenance dose 75 mg/day
  Interventions: Drug: Clopidogrel
- Prasugrel 30/5 Low Weight/Elderly (Experimental): Loading dose 30 mg followed by maintenance dose 5 mg/day
  Interventions: Drug: Prasugrel
- Clopidogrel 300/75 Low Weight/Elderly (Active Comparator): Loading dose 300 mg followed by maintenance dose 75 mg/day
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Oral, daily, 90 days
  Other Names: LY640315; Effient; Efient; CS-747
  Arms: Prasugrel 30/5 Low Weight/Elderly; Prasugrel 30/5 Primary; Prasugrel 30/7.5 Primary; Prasugrel 60/10 Primary
Drug: Clopidogrel — Oral, daily, 90 days
  Other Names: Plavix
  Arms: Clopidogrel 300/75 Low Weight/Elderly; Clopidogrel 300/75 Primary

SUMMARY:
The study will compare the safety and efficacy of prasugrel, administered at different doses with clopidogrel in the treatment of Asian participants with acute coronary syndrome (ACS) undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* A person who has been diagnosed with acute coronary syndrome (ACS) and is to undergo a percutaneous coronary intervention (PCI)
* A person who is of East or Southeast Asian descent
* A person who is of the legal age of 18 (or age 21 in Singapore) and is mentally competent to provide a signed written informed consent before entering the study
* If a woman is of childbearing potential, she must test negative for pregnancy and agree to use a reliable method of birth control

Exclusion Criteria:

* A person who has a severe cardiovascular condition such as cardiogenic shock at the time of randomization, ventricular arrhythmias or congestive heart failure
* A person who is at an increased risk of bleeding (e.g. active internal bleeding, history of bleeding disorder, recent fibrinolytic therapy before randomization into the study)
* A person who has prior history of any one of the following: ischemic or hemorrhagic stroke; intracranial neoplasm, arteriovenous malformation, or aneurysm; prior history of transient ischemic attack (TIA)
* A person who needs to take other antiplatelet therapy other than Aspirin for the duration of the study
* A person who receives daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX2) inhibitors that cannot be discontinued
* A person who has a severe liver disease, such as cirrhosis
* A person who has a condition such as alcoholism, mental illness, or drug dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- China (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District
- Thailand (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangkok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiang Mai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 4 treatment arms and had 2 cohorts; a Primary Cohort (≥60 kilograms [kg] and age <75 years) and a Low Weight/Elderly cohort (<60 kg or age ≥75 years). Randomization was stratified by country, cohort and anticipated glycoprotein (GP) IIb/IIIa inhibitor use.
Pre-assignment Details: One participant who was enrolled based on weight >60 kg was not assigned to primary cohort due to no weight entered in case report form.
  Low Weight/Elderly Cohort was only assigned to prasugrel 30-mg loading dose (LD)/5-mg maintenance dose (MD) or clopidogrel 300-mg LD/75-mg MD due to evidence of increased bleeding risk for these populations.
Groups:
- Prasugrel 60/10 Primary: Population includes participants randomly assigned to receive prasugrel 60-mg loading dose (LD) followed by prasugrel 10-mg maintenance dose (MD) daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/7.5 Primary: Population includes participants randomly assigned to receive prasugrel 30-mg LD followed by prasugrel 7.5-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/5 Primary: Population includes participants randomly assigned to receive prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Clopidogrel 300/75 Primary: Population includes participants randomly assigned to receive clopidogrel 300-mg LD followed by prasugrel 75-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/5 Low Weight/Elderly: Population includes participants randomly assigned to receive prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the Low Weight/Elderly cohort (participant weight <60 kg or age ≥75 years)
- Clopidogrel 300/75 Low Weight/Elderly: Population includes participants randomly assigned to receive clopidogrel 300-mg LD followed by prasugrel 75-mg MD daily in the Low Weight/Elderly cohort (participant weight <60 kg or age ≥75 years)
Period: Overall Study
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Started | 124 (Number of participants "STARTED" equals the number of participants randomized.) | 124 | 137 | 138 | 96 | 100 (Total 720 participants were randomized; 1 was not included in a cohort as baseline weight missing.)
Received at Least 1 Dose of Study Drug | 117 (Baseline Characteristics (below) include those who received ≥1 dose study drug, not all who STARTED.) | 122 | 133 | 135 | 91 | 93
Completed | 91 | 96 | 108 | 106 | 64 (6 participants not completed due to death; 1 additional death occurred after study discontinuation.) | 63
Not Completed | 33 | 28 | 29 | 32 | 32 | 37
Not completed — Death | 5 | 4 | 3 | 2 | 6 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 19 | 19 | 18 | 23 | 16 | 21
Not completed — Sponsor Decision | 1 | 2 | 3 | 4 | 5 | 7
Not completed — No study drug received | 7 | 2 | 4 | 3 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel 60/10 Primary: Study treatment of prasugrel 60-mg LD followed by prasugrel 10-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
  Reporting groups for Baseline Characteristics do not include all randomized participants (n=720), but includes all randomized participants who received at least 1 dose of study drug.
- Prasugrel 30/7.5 Primary: Study treatment of prasugrel 30-mg LD followed by prasugrel 7.5-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/5 Primary: Study treatment of prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Clopidogrel 300/75 Primary: Study treatment of clopidogrel 300-mg LD followed by clopidogrel 75-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/5 Low Weight/Elderly: Study treatment of prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the Low Weight/Elderly cohort (participant weight <60 kg or age ≥75 years)
- Clopidogrel 300/75 Low Weight/Elderly: Study treatment of clopidogrel 300-mg LD followed by clopidogrel 75-mg MD daily in the Low Weight/Elderly cohort (participant weight <60 kg or age ≥75 years)
- Total: Total of all reporting groups
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly | Total
Number analyzed (Participants) | 117 | 122 | 133 | 135 | 91 | 93 | 691
Age Continuous [Mean (Standard Deviation); unit: years] — Total mean age is based on all randomized participants who received at least 1 dose of study drug, and for whom information was available (n=689).
  years
    Mean Age Overall | 58.3 (9.83) | 57.7 (9.47) | 57.2 (10.49) | 58.3 (8.95) | 68.5 (9.74) | 69.1 (12.08) | 60.8 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 27 | 24 | 45 | 48 | 174
  Male | 101 | 108 | 106 | 111 | 46 | 45 | 517
Region of Enrollment [Number; unit: participants]
  China | 85 | 85 | 93 | 95 | 64 | 61 | 483
  Korea, Republic of | 15 | 19 | 20 | 19 | 13 | 15 | 101
  Taiwan | 12 | 14 | 15 | 16 | 10 | 11 | 78
  Thailand | 5 | 4 | 5 | 5 | 4 | 6 | 29
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m²)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m²)
    BMI | 25.86 (2.907) | 25.75 (2.990) | 26.06 (2.637) | 26.19 (2.999) | 22.02 (4.106) | 22.10 (3.166) | 24.74 (3.510)
Qualifying Diagnosis [Number; unit: participants]
  Unstable angina (UA) | 32 | 42 | 38 | 41 | 26 | 30 | 209
  Non-ST segment elevation myocardial infarction | 13 | 16 | 21 | 17 | 10 | 10 | 87
  ST segment elevation myocardial infarction | 72 | 64 | 74 | 77 | 55 | 53 | 395

OUTCOME MEASURES:

1. Primary Outcome: Adenosine Diphosphate (ADP)-Induced P2Y12 Receptor-mediated Platelet Aggregation (P2Y12 Reaction Units; PRU) Using the Accumetrics VerifyNow (VN) P2Y12 Assay at 4 Hours Post-Loading Dose (LD) in Primary Cohort (≥60 kg and <75 Years)
Description: ADP-induced PRU represents the rate and extent of ADP-stimulated platelet aggregation and serves as a biomarker of clinical efficacy, with lower values indicating greater P2Y12 platelet inhibition.
  Observed PRU values are presented with statistical comparisons of difference in least squares mean (LS mean) PRU values between prasugrel and clopidogrel.
  Efficacy analyses are analyzed and presented separately for the LD and maintenance dose (MD) phase.
Time Frame: At 4 hours following LD administration
Population: Per Protocol Set (PPS) LD population
  PPS: all randomized participants with ≥1 dose study drug, ≥1 post-baseline platelet aggregation measurement, no significant protocol violations
  LD population: never used glycoprotein (GP) IIb/IIIa inhibitor during index hospitalization and received percutaneous coronary intervention (PCI) for index event
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Prasugrel 60-mg LD Primary: Population includes participants in primary cohort randomly assigned to receive prasugrel 60-mg LD
- Prasugrel 30-mg LD Primary: Population includes participants in primary cohort who were randomly assigned to receive a prasugrel 30-mg LD (including participants in both Prasugrel 30/7.5 Primary and Prasugrel 30/5 Primary populations).
- Clopidogrel 300-mg LD Primary: Population includes participants in primary cohort who were randomly assigned to receive a clopidogrel 300-mg LD.
Arm/Group | Prasugrel 60-mg LD Primary | Prasugrel 30-mg LD Primary | Clopidogrel 300-mg LD Primary
Number analyzed (Participants) | 35 | 79 | 44
PRU | 88.5 (104.86) | 124.2 (117.28) | 261.8 (83.87)
Statistical Analysis 1: Comparison: Prasugrel 60-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Linear mixed effects model: treatment, visit, treatment-by-visit interaction, gender, country as fixed effects, baseline PRU as covariate, participant as random effect was used. Difference in PRU = prasugrel - clopidogrel; Kenward-Roger method was used to estimate denominator degrees of freedom for fixed effects. Invalid measurements excluded; Least Square (LS) Mean Difference in PRU = -183, 95% CI 2-sided [-229 to -137]
Statistical Analysis 2: Comparison: Prasugrel 30-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference in PRU = -139, 95% CI 2-sided [-177 to -102]

2. Secondary Outcome: Adenosine Diphosphate (ADP)-Induced P2Y12 Reaction Units (PRU) Using the Accumetrics VerifyNow (VN) P2Y12 Assay at 30 Minutes, 2 and 4 Hours Post-Loading Dose (LD) in Primary (≥60 kg and <75 Years) and Low Weight/Elderly (<60 kg or ≥75 Years) Cohorts.
Description: Efficacy analyses analyzed and presented separately for LD and maintenance dose (MD) phase. Analysis compares PRU for prasugrel LDs (30 mg and 60 mg) with clopidogrel 300-mg LD at 30 minutes post-LD.
  Data for Primary Cohort at 4 hours post-LD, already presented in first Primary Outcome Measure, are also presented here.
  ADP-induced PRU serves as biomarker of clinical efficacy, with lower values indicating greater P2Y12 platelet inhibition.
  Observed PRU values presented with statistical comparisons of least-squares mean (LS mean) difference between prasugrel and clopidogrel.
Time Frame: At 30 minutes, 2 hours, and 4 hours following LD administration
Population: Per Protocol Set (PPS) LD population PPS: all randomized participants with at least 1 dose study drug, ≥1 post-baseline platelet aggregation measurement, no significant protocol violations
  LD population: never used glycoprotein (GP)IIb/IIIa inhibitor during index hospitalization, received percutaneous coronary intervention (PCI) for index event
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Prasugrel 30-mg LD Low Weight/Elderly: Population includes participants in low weight/elderly cohort who were randomly assigned to receive a prasugrel 30-mg LD.
- Clopidogrel 300-mg LD Low Weight/Elderly: Population includes participants in low weight/elderly cohort who randomly assigned to receive a clopidogrel 300-mg LD.
Arm/Group | Prasugrel 60-mg LD Primary | Prasugrel 30-mg LD Primary | Clopidogrel 300-mg LD Primary | Prasugrel 30-mg LD Low Weight/Elderly | Clopidogrel 300-mg LD Low Weight/Elderly
Number analyzed (Participants) | 43 | 90 | 54 | 33 | 34
PRU
  30 min (n=40, n=79, n=48, n=33, n=34) | 250.5 (109.02) | 280.4 (112.58) | 312.1 (72.41) | 311.2 (96.46) | 379.5 (53.29)
  2 hours (n=37, n=80, n=49, n=33, n=33) | 116.9 (116.48) | 178.8 (128.37) | 289.5 (71.77) | 171.8 (123.37) | 339.0 (74.03)
  4 hours (n=35, n=79, n=44, n=33, n=33) | 88.5 (104.86) | 124.2 (117.28) | 261.8 (83.87) | 127.3 (106.38) | 337.8 (85.15)
Statistical Analysis 1: Comparison: Prasugrel 60-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p = 0.0058, Mixed Models Analysis — P-value for 30 minutes post-LD Linear mixed effects model: treatment, visit, treatment-by-visit interaction, gender, country as fixed effects, baseline PRU as covariate, participant as random effect Difference in PRU = prasugrel - clopidogrel; Kenward-Roger method was used to estimate the denominator degrees of freedom for fixed effects. Invalid measurements were excluded; LS mean difference in PRU = -57, 95% CI 2-sided [-97 to -17]
Statistical Analysis 2: Comparison: Prasugrel 30-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p = 0.0365, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -35, 95% CI 2-sided [-68 to -2]
Statistical Analysis 3: Comparison: Prasugrel 30-mg LD Low Weight/Elderly vs Clopidogrel 300-mg LD Low Weight/Elderly; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -68, 95% CI 2-sided [-104 to -32]
Statistical Analysis 4: Comparison: Prasugrel 60-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 2 hours post-LD Linear mixed effects model: treatment, visit, treatment-by-visit interaction, gender, country as fixed effects, baseline PRU as covariate, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -160, 95% CI 2-sided [-211 to -110]
Statistical Analysis 5: Comparison: Prasugrel 30-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 4]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -115, 95% CI 2-sided [-156 to -73]
Statistical Analysis 6: Comparison: Prasugrel 30-mg LD Low Weight/Elderly vs Clopidogrel 300-mg LD Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 4]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -171, 95% CI 2-sided [-216 to -125]
Statistical Analysis 7: Comparison: Prasugrel 30-mg LD Low Weight/Elderly vs Clopidogrel 300-mg LD Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 4 hours post-LD Linear mixed effects model: treatment, visit, treatment-by-visit interaction, gender, country as fixed effects, baseline PRU as covariate, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -212, 95% CI 2-sided [-259 to -167]

3. Secondary Outcome: Adenosine Diphosphate (ADP)-Induced P2Y12 Reaction Units (PRU) Using the Accumetrics VerifyNow (VN) P2Y12 Assay at During Maintenance Dose (MD) Phase at 30 Days and 90 Days in Primary Cohort and Low Weight/Elderly Cohort
Description: Efficacy analyses analyzed and presented separately for loading dose (LD) and MD phase. Analysis compares PRU for 3 prasugrel MDs (10 mg, 7.5 mg, and 5 mg) with clopidogrel 75-mg MD at 30 days post-MD.
  Data for Primary Cohort at 30 days post-LD, already presented in second Primary Outcome Measure, are also presented here.
  ADP-induced PRU serves as a biomarker of clinical efficacy, with lower values indicating greater P2Y12 platelet inhibition.
  Observed PRU values are presented with statistical comparisons of least squares (LS) mean difference between prasugrel and clopidogrel.
Time Frame: At 30 Days and 90 days during MD therapy
Population: Per Protocol Set (PPS) MD population PPS: all randomized participants who had at least 1 dose of study drug, ≥1 post-baseline platelet aggregation measurement, and no significant protocol violations in MD population: received percutaneous coronary intervention (PCI) for index event
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 74 | 69 | 75 | 89 | 55 | 54
PRU
  30 days (n=69, n=63, n=69, n=78, n=47, n=48) | 71.6 (65.56) | 99.3 (72.63) | 150.8 (77.76) | 206.5 (72.68) | 134.2 (80.29) | 237.5 (108.32)
  90 Days (n=60, n=57, n=64, n=72, n=43, n=42) | 64.8 (55.99) | 89.4 (91.75) | 138.5 (80.42) | 188.3 (81.24) | 128.5 (70.42) | 219.6 (95.06)
Statistical Analysis 1: Comparison: Prasugrel 30/5 Low Weight/Elderly vs Clopidogrel 300/75 Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, LS Mean Difference in PRU — P-value for 30 days. A linear mixed effects model including treatment, visit, treatment-by-visit interaction, gender, country as fixed effects, baseline PRU as covariate, participant as random effect Difference in PRU was prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in PRU = -119, 95% CI 2-sided [-166 to -73]
Statistical Analysis 2: Comparison: Prasugrel 60/10 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 90 days. A linear mixed effects model including treatment, visit, treatment-by-visit interaction, gender, country as fixed effects, baseline PRU as covariate, participant as random effect Difference in PRU was prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in PRU = -113, 95% CI 2-sided [-154 to -73]
Statistical Analysis 3: Comparison: Prasugrel 30/7.5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in PRU = -85, 95% CI 2-sided [-121 to -48]
Statistical Analysis 4: Comparison: Prasugrel 30/5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.0647, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in PRU = -35, 95% CI 2-sided [-72 to 2]
Statistical Analysis 5: Comparison: Prasugrel 30/5 Low Weight/Elderly vs Clopidogrel 300/75 Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in PRU = -100, 95% CI 2-sided [-143 to -57]

4. Secondary Outcome: Percent Inhibition of Adenosine Diphosphate (ADP)-Induced P2Y12 Reaction Units (PRU) at 30 Minutes, 2 Hours, and 4 Hours Post-Loading Dose (LD) in Primary in Primary Cohort and Low Weight/Elderly Cohort
Description: A higher percentage (percent inhibition least squares mean [LS mean]) represents greater platelet inhibition.
Time Frame: 30 minutes, 2 hours, and 4 hours following LD administration
Population: Per Protocol Set (PPS) LD population PPS: all randomized participants with at least 1 dose study drug, ≥1 post-baseline platelet aggregation measurement, no significant protocol violations LD population: never used glycoprotein (GP) IIb/IIIa inhibitor during index hospitalization, received percutaneous coronary intervention (PCI) for index event
Measure: Number; unit: Percent inhibition
Groups:
- Prasugrel 60-mg LD Primary: Population includes participants in primary cohort who were treated with a prasugrel 60-mg LD.
- Prasugrel 30-mg LD Primary: Population includes participants in primary cohort who were treated with a prasugrel 30-mg LD(including participants in both Prasugrel 30/7.5 Primary and Prasugrel 30/5 Primary populations).
- Clopidogrel 300-mg LD Primary: Population includes participants in primary cohort who were treated with a clopidogrel 300-mg LD.
- Prasugrel 30-mg LD Low Weight/Elderly: Population includes participants in low weight/elderly cohort who were treated with a prasugrel 30-mg LD.
- Clopidogrel 300-mg LD Low Weight/Elderly: Population includes participants in low weight/elderly cohort who were treated with a clopidogrel 300-mg LD.
Arm/Group | Prasugrel 60-mg LD Primary | Prasugrel 30-mg LD Primary | Clopidogrel 300-mg LD Primary | Prasugrel 30-mg LD Low Weight/Elderly | Clopidogrel 300-mg LD Low Weight/Elderly
Number analyzed (Participants) | 43 | 90 | 54 | 33 | 34
Percent inhibition
  30 minutes (n=40, n=79, n=47, n=32, n=31) | 10 | 4 | -5 | 11 | 0
  2 hours (n=37, n=80, n=48, n=33, n=33) | 49 | 34 | -2 | 51 | 2
  4 hours (n=34, n=79, n=43, n=33, n=33) | 65 | 51 | 4 | 63 | 7
Statistical Analysis 1: Comparison: Prasugrel 60-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p = 0.0072, Mixed Models Analysis — P-value for 30 minutes post-LD Linear mixed effects model: treatment, visit (0.5 hours to 4 hours), treatment-by-visit interaction, gender, country as fixed effects, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 15, 95% CI 2-sided [4 to 27]
Statistical Analysis 2: Comparison: Prasugrel 30-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p = 0.0647, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 9, 95% CI 2-sided [-1 to 18]
Statistical Analysis 3: Comparison: Prasugrel 30-mg LD Low Weight/Elderly vs Clopidogrel 300-mg LD Low Weight/Elderly; Test type: Superiority or Other; p = 0.0054, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 11, 95% CI 2-sided [3 to 19]
Statistical Analysis 4: Comparison: Prasugrel 60-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 2 hours post-LD Linear mixed effects model: treatment, visit (0.5 hours to 4 hours), treatment-by-visit interaction, gender, country as fixed effects, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 51, 95% CI 2-sided [36 to 66]
Statistical Analysis 5: Comparison: Prasugrel 30-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 4]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 36, 95% CI 2-sided [23 to 48]
Statistical Analysis 6: Comparison: Prasugrel 30-mg LD Low Weight/Elderly vs Clopidogrel 300-mg LD Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 4]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 49, 95% CI 2-sided [36 to 61]
Statistical Analysis 7: Comparison: Prasugrel 60-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 4 hours post-LD Linear mixed effects model: treatment, visit (0.5 hours to 4 hours), treatment-by-visit interaction, gender, country as fixed effects, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 62, 95% CI 2-sided [47 to 76]
Statistical Analysis 8: Comparison: Prasugrel 30-mg LD Primary vs Clopidogrel 300-mg LD Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 7]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 48, 95% CI 2-sided [36 to 59]
Statistical Analysis 9: Comparison: Prasugrel 30-mg LD Low Weight/Elderly vs Clopidogrel 300-mg LD Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 7]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 56, 95% CI 2-sided [44 to 68]

5. Secondary Outcome: Percent Inhibition of Adenosine Diphosphate (ADP)-Induced P2Y12 Reaction Units (PRU) During the Maintenance Dose (MD) Phase at 30 Days and 90 Days in Primary Cohort and Low Weight/Elderly Cohort
Description: A higher percentage (percent inhibition least squares mean [LS mean]) represents greater platelet inhibition.
Time Frame: 30 days and at 90 days during MD therapy
Population: Per Protocol Set (PPS) MD population
  PPS: all randomized participants who had at least 1 dose of study drug, ≥1 post-baseline platelet aggregation measurement, and no significant protocol violations
  MD population: received percutaneous coronary intervention (PCI) for index event
Measure: Number; unit: Percent inhibition
Groups:
- Prasugrel 60/10 Primary: Population includes participants randomly assigned to receive prasugrel 60-mg LD followed by prasugrel 10-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Clopidogrel 300/75 Primary: Population includes participants randomly assigned to receive clopidogrel 300-mg LD followed by clopidogrel 75-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Clopidogrel 300/75 Low Weight/Elderly: Population includes participants randomly assigned to receive clopidogrel 300-mg LD followed by clopidogrel 75-mg MD daily in the low weight/elderly cohort (participant weight <60 kg or age ≥75 years)
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 74 | 69 | 75 | 89 | 55 | 54
Percent inhibition
  30 Days (n=69, n=63, n=68, n=78, n=47, n=48) | 67 | 60 | 45 | 29 | 68 | 32
  90 Days (n=60, n=57, n=64, n=72, n=43, n=42) | 73 | 66 | 48 | 38 | 69 | 38
Statistical Analysis 1: Comparison: Prasugrel 60/10 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 30 days post-LD Linear mixed effects model: treatment, visit (30, 90 days during MD), treatment-by-visit interaction, gender, country as fixed effects, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 38, 95% CI 2-sided [27 to 50]
Statistical Analysis 2: Comparison: Prasugrel 30/7.5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 32, 95% CI 2-sided [21 to 42]
Statistical Analysis 3: Comparison: Prasugrel 30/5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 17, 95% CI 2-sided [6 to 28]
Statistical Analysis 4: Comparison: Prasugrel 30/5 Low Weight/Elderly vs Clopidogrel 300/75 Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 37, 95% CI 2-sided [24 to 50]
Statistical Analysis 5: Comparison: Prasugrel 60/10 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — P-value for 90 days post-LD Linear mixed effects model: treatment, visit (30, 90 days during MD), treatment-by-visit interaction, gender, country as fixed effects, participant as random effect Difference in PRU = prasugrel - clopidogrel; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 35, 95% CI 2-sided [18 to 52]
Statistical Analysis 6: Comparison: Prasugrel 30/7.5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 5]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 28, 95% CI 2-sided [13 to 44]
Statistical Analysis 7: Comparison: Prasugrel 30/5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.1898, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 5]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 11, 95% CI 2-sided [-5 to 27]
Statistical Analysis 8: Comparison: Prasugrel 30/5 Low Weight/Elderly vs Clopidogrel 300/75 Low Weight/Elderly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 5]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference in Percent Inhibition = 32, 95% CI 2-sided [18 to 45]

6. Secondary Outcome: Summary of Myocardial Infarction (MI), Stroke, Stent Thrombosis and Urgent Target Vessel Revascularization (UTVR) in Primary Cohort and Low Weight/Elderly Cohort
Description: Nonfatal MI: American College of Cardiology (ACC) definition Nonfatal stroke: rapid onset of new, persistent neurologic deficit lasting >24 hours; classified as either ischemic or hemorrhagic based on imaging data, if available, or uncertain cause if imaging data was not available.
  Stent thrombosis: defined as definite, probable, or possible, based on Academic Research Consortium definitions.
  UTVR: percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) for recurrent ischemia. Revascularization must have included the vessel(s) dilated at the initial procedure
Time Frame: Randomization through end of study (90 days)
Population: Full analysis set (FAS)
  FAS: all randomized subjects who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 117 | 122 | 133 | 136 | 91 | 93
Participants
  Fatal MI | 1 | 0 | 0 | 0 | 1 | 0
  Nonfatal MI | 1 | 0 | 1 | 1 | 0 | 2
  Fatal Stroke | 0 | 1 | 0 | 0 | 0 | 0
  Nonfatal Stroke | 0 | 1 | 0 | 0 | 2 | 0
  Definite Stent Thrombosis | 0 | 1 | 0 | 1 | 1 | 0
  UTVR | 1 | 1 | 0 | 1 | 1 | 1

7. Primary Outcome: Adenosine Diphosphate (ADP)-Induced P2Y12 Reaction Units (PRU) Using the Accumetrics VerifyNow (VN) P2Y12 Assay at 30 Days During Maintenance Dose (MD) Administration in Primary Cohort
Description: Efficacy analyses are analyzed and presented separately for the loading dose (LD) and MD phase. This primary outcome analysis compares PRU for the 3 prasugrel MDs (10 mg, 7.5 mg, and 5 mg) with the clopidogrel 75-mg MD at 30 days post-MD in the primary cohort (participants who weighed ≥60 kg and were <75 years).
  ADP-induced PRU serves as a biomarker of clinical efficacy, with lower values indicating greater P2Y12 platelet inhibition.
  Observed PRU values are presented with statistical comparisons of LS mean difference between prasugrel and clopidogrel.
Time Frame: At 30 days during MD therapy
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Prasugrel 60/10 Primary: Population includes participants in primary cohort randomly assigned to receive prasugrel 60-mg LD followed by prasugrel 10-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/7.5 Primary: Population includes participants in primary cohort randomly assigned to receive prasugrel 30-mg LD followed by prasugrel 7.5-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Prasugrel 30/5 Primary: Population includes participants in primary cohort randomly assigned to receive prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the primary cohort (participant weight ≥60 kg and age <75 years)
- Clopidogrel 300/75 Primary: Population includes participants in primary cohort randomly assigned to receive clopidogrel 300-mg LD followed by clopidogrel 75-mg MD daily in the primary cohort participant weight ≥60 kg and age <75 years)
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary
Number analyzed (Participants) | 69 | 63 | 69 | 78
PRU | 71.6 (65.56) | 99.3 (72.63) | 150.8 (77.76) | 206.5 (72.68)
Statistical Analysis 1: Comparison: Prasugrel 60/10 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -110, 95% CI 2-sided [-143 to -76]
Statistical Analysis 2: Comparison: Prasugrel 30/7.5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -92, 95% CI 2-sided [-123 to -60]
Statistical Analysis 3: Comparison: Prasugrel 30/5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS mean difference in PRU = -51, 95% CI 2-sided [-83 to -19]

8. Secondary Outcome: Risk of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), or Non-fatal Stroke
Description: Risk was defined as the number of participants with events of CV death, nonfatal MI, or nonfatal stroke.
  CV death: death caused by CV event or not clearly attributable to non-CV causes.
  Nonfatal MI: per adapted American College of Cardiology definition.
  Nonfatal stroke: rapid onset of new, persistent neurologic deficit lasting more than 24 hours; either ischemic or hemorrhagic based on imaging data, if available, or uncertain cause if imaging data was not available.
  As a consequence of the overall low number of reported clinical events, composite endpoints were not analyzed.
Time Frame: 30 days and 90 days
Population: As a consequence of the overall low number of reported clinical events, composite endpoints were not analyzed; thus zero participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Risk of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), or Urgent Target Vessel Revascularization (UTVR)
Description: Risk was defined as the number of participants with events of CV death, nonfatal MI, or UTVR.
  UTVR: percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) for recurrent ischemia. Revascularization must have included the vessel(s) dilated at the initial procedure.
  As a consequence of the overall low number of reported clinical events, composite endpoints were not analyzed.
Time Frame: 30 days and 90 days
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Risk of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, or Recurrent Myocardial Ischemia Requiring Hospitalization
Description: Risk was defined as the number of events of CV death, nonfatal MI, nonfatal stroke or recurrent myocardial ischemia requiring hospitalization.
  Recurrent myocardial ischemia requiring hospitalization: rehospitalization for symptoms of myocardial ischemia at rest with either new ST-segment deviation ≥1 mm, or performance of a coronary revascularization procedure percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) during the same hospital stay.
  As a consequence of the overall low number of reported clinical events, composite endpoints were not analyzed.
Time Frame: 30 days and 90 days
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Risk of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, Urgent Target Vessel Revascularization (UTVR), or Recurrent Myocardial Ischemia Requiring Hospitalization (Analyzed Individually)
Description: Risk was defined as the number of participants with events of CV death, nonfatal MI, nonfatal stroke, UTVR, or recurrent myocardial ischemia requiring hospitalization.
Time Frame: 30 days and 90 days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Risk of Definite or Probable Stent Thrombosis Per ARC (Academic Research Consortium) Definition
Description: Risk was defined as the number of participants with events of definite or probable stent thrombosis.
  As a consequence of the overall low number of reported clinical events, composite endpoints were not analyzed.
Time Frame: 30 days and 90 days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Risk of Definite, Probable, or Possible Stent Thrombosis Per Academic Research Consortium (ARC) Definition
Description: Risk was defined as the number of participants with events of definite, probable, or possible stent thrombosis.
  As a consequence of the overall low number of reported clinical events, composite endpoints were not analyzed.
Time Frame: 90 days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Risk of All-cause Death in Primary Cohort and Low Weight/Elderly Cohort
Description: Risk was defined as the number of participants with events of all-cause death.
Time Frame: Randomization through end of study (90 days)
Population: Full Analysis Set (FAS): all randomized subjects who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 117 | 122 | 133 | 135 | 91 | 93
Participants | 5 | 4 | 3 | 2 | 7 | 1
Statistical Analysis 1: Comparison: Prasugrel 60/10 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.255, Fisher Exact
Statistical Analysis 2: Comparison: Prasugrel 30/7.5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.427, Fisher Exact
Statistical Analysis 3: Comparison: Prasugrel 30/5 Primary vs Clopidogrel 300/75 Primary; Test type: Superiority or Other; p = 0.683, Fisher Exact
Statistical Analysis 4: Comparison: Prasugrel 30/5 Low Weight/Elderly vs Clopidogrel 300/75 Low Weight/Elderly; Test type: Superiority or Other; p = 0.034, Fisher Exact

15. Secondary Outcome: Incidence of Non-coronary Artery Bypass Graft (CABG) Related Thrombolysis in Myocardial Infarction (TIMI) Life-threatening (a Subset of Non-CABG-related TIMI Major Bleeding), Major, Minor, and Minimal Bleeding
Description: Bleeding events were classified and analyzed in accordance with the TIMI criteria definitions.
  Major bleeding: any intracranial hemorrhage (ICR) OR any clinically overt bleeding (including bleeding evident on imaging studies) associated with a fall in hemoglobin (Hgb) of ≥5 grams/deciliter (gm/dL) from baseline.
  Minor bleeding: any clinically overt bleeding associated with a fall in Hgb of ≥3 but <5 gm/dL from baseline.
  Insignificant bleeding: any bleeding event that does not meet criteria for a Major or Minor bleed.
Time Frame: Randomization through end of study (90 days)
Population: Safety analysis set (SAS): all randomized participants with at least 1 dose of study drug
  Two (2) participants had no event date; time from start of therapy to event was missing and thus they were not included in this table.
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 117 | 122 | 133 | 136 | 91 | 93
participants
  ≤3 Days of LD Major | 2 | 0 | 0 | 0 | 2 | 2
  ≤3 Days of LD Life Threatening | 2 | 0 | 0 | 0 | 2 | 1
  ≤3 Days of LD Minor | 1 | 0 | 2 | 1 | 1 | 0
  ≤3 Days of LD Minimal | 5 | 4 | 6 | 4 | 1 | 1
  >3 Days of LD Major | 2 | 1 | 0 | 0 | 1 | 2
  >3 Days of LD Life Threatening | 0 | 1 | 0 | 0 | 1 | 0
  >3 Days of LD Minor | 0 | 0 | 0 | 0 | 0 | 2
  >3 Days of LD Minimal | 1 | 2 | 7 | 3 | 2 | 3

16. Secondary Outcome: Incidence of CABG-related TIMI Major or Minor Bleeding.
Time Frame: Randomization through end of study (90 days)
Population: Safety Analysis Set (SAS): all randomized participants with at least 1 dose of study drug
  In 10 participants, study drug discontinued due to planned CABG. 1 participant had CABG reported on revascularization case report form (CRF); no reports of CABG bleeding event
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 117 | 122 | 133 | 136 | 91 | 93
participants | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Inpatient Healthcare Resource Utilization
Description: Healthcare resource utilization data were modeled from historical analyses to determine initial hospitalization costs, total 30-day medical care costs, and total 90-day medical care costs.
Time Frame: Initial hospitalization, 30 days, 90 days
Population: As a consequence of the overall low number of reported clinical events, inpatient healthcare resource utilization data were not analyzed; thus zero participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Genetic Variation Related to Drug Metabolism and Transport Substudy Result Summary
Description: The primary hypothesis for the genetics substudy was that CYP2C19 genetic variation has a significant effect on pharmacodynamic (PD) response to clopidogrel but not on PD response to prasugrel per change in PRU as measured by the Accumetrics VerifyNow P2Y12 device.
  Participants were classified by CYP2C19 genotype into predicted metabolic phenotypes according to literature-based functional predictions. These classifications were clustered into 2 groups: extensive metabolizer (EM) and reduced metabolizer (RM).
  A higher value for change in PRU indicates a greater level of platelet inhibition.
Time Frame: Baseline to 4 hours post-loading dose (LD), 30 days and 90 days during maintenance dose (MD) phase
Population: Pharmacodynamic analysis set is subset of FAS (≥1 genetics sample, ≥1 dose of study drug, ≥1 post-baseline PRU measurement, no significant protocol violations). Genetics subset LD population never used glycoprotein (GP) IIb/IIIa inhibitor during index hospitalization.
  Participants classified as EM or RM. Invalid measurements of PRU were excluded.
Measure: Mean (Standard Deviation); unit: Change in PRU
Groups:
- Prasugrel 60/10 PD: Population includes participants in genetics substudy who were randomly assigned to receive a prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the Primary Cohort.
- Prasugrel 30/7.5 PD: Population includes participants in genetics substudy who were randomly assigned to receive a prasugrel 30-mg LD followed by prasugrel 7.5-mg MD daily in the Primary and Low Weight/Elderly Cohorts combined.
- Prasugrel 30/5 PD: Population includes participants in genetics substudy who were randomly assigned to receive a prasugrel 30-mg LD followed by prasugrel 5-mg MD daily in the Primary and Low Weight/Elderly Cohorts combined.
- Clopidogrel 300/75 PD: Population includes participants in genetics substudy who were randomly assigned to receive a clopidogrel 300-mg LD followed by clopidogrel 75-mg MD daily in the Primary and Low Weight/Elderly Cohorts combined.
Arm/Group | Prasugrel 60/10 PD | Prasugrel 30/7.5 PD | Prasugrel 30/5 PD | Clopidogrel 300/75 PD
Number analyzed (Participants) | 83 | 76 | 155 | 162
Change in PRU
  4 hours, EM (n=15, n=18, n=27, n=31) | -162.9 (154.30) [-397 to 144] | -198.8 (90.71) [-230 to 215] | -217.2 (83.52) | -9.7 (72.30)
  4 hours, RM (n=18, n=21, n=45, n=45) | -245.9 (102.77) | -183.3 (123.29) | -181.9 (129.47) | -22.2 (72.84)
  30 days, EM (n=17, n=21, n=31, n=30) | -193.9 (98.17) | -196.5 (88.90) | -187.5 (94.79) | -110.6 (83.49)
  30 days, RM (n=19, n=21. n=43, n=47) | -250.3 (90.17) | -208.5 (74.23) | -152.8 (88.97) | -81.7 (70.56)
  90 days, EM (n=12, n=18, n=30, n=28) | -203.8 (102.89) | -210.0 (110.68) | -187.2 (92.70) | -141.0 (75.58)
  90 days, RM (n=17, n=21, n=36, n=41) | -267.5 (70.86) | -225.7 (76.52) | -164.1 (75.90) | -100.7 (92.24)

19. Secondary Outcome: Risk of CV Death, Nonfatal MI, Nonfatal Stroke, UTVR, or Recurrent Myocardial Ischemia Requiring Hospitalization (Analyzed Individually)
Description: Risk of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, Urgent Target Vessel Revascularization (UTVR), or Recurrent Myocardial Ischemia Requiring Hospitalization (Analyzed Individually)
Time Frame: 30 days and 90 days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Prasugrel 60/10 Primary: Primary = participant weight ≥60 kg and age <75 years. Loading dose 60 mg followed by maintenance dose 10 mg/day.
- Prasugrel 30/7.5 Primary: Primary = participant weight ≥60 kg and age <75 years. Loading dose 30mg followed by maintenance dose 7.5 mg/day
- Prasugrel 30/5 Primary: Primary = participant weight ≥60 kg and age <75 years. Loading dose 30 mg followed by maintenance dose 5 mg/day.
- Clopidogrel 300/75 Primary: Primary = participant weight ≥60 kg and age <75 years. Loading dose 300 mg followed by maintenance dose 75 mg/day
- Prasugrel 30/5 Low Weight/Elderly: Low Weight/Elderly = participant weight <60 kg or age ≥75 years. Loading dose 30 mg followed by maintenance dose 5 mg/day.
- Clopidogrel 300/75 Low Weight/Elderly: Low Weight/Elderly = participant weight <60 kg or age ≥75 years. Loading dose 300 mg followed by maintenance dose 75 mg/day
- Clopidogrel 300/75 No Weight: Participant didn't have weight recorded. Loading dose 300 mg followed by maintenance dose 75 mg/day
Arm/Group | Prasugrel 60/10 Primary | Prasugrel 30/7.5 Primary | Prasugrel 30/5 Primary | Clopidogrel 300/75 Primary | Prasugrel 30/5 Low Weight/Elderly | Clopidogrel 300/75 Low Weight/Elderly | Clopidogrel 300/75 No Weight
Serious Adverse Events (participants affected / at risk) | 8/117 | 7/122 | 4/133 | 6/135 | 9/91 | 10/93 | 0/1
Other Adverse Events (participants affected / at risk) | 54/117 | 38/122 | 45/133 | 49/135 | 28/91 | 34/93 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel 60/10 Primary (N=117) | Prasugrel 30/7.5 Primary (N=122) | Prasugrel 30/5 Primary (N=133) | Clopidogrel 300/75 Primary (N=135) | Prasugrel 30/5 Low Weight/Elderly (N=91) | Clopidogrel 300/75 Low Weight/Elderly (N=93) | Clopidogrel 300/75 No Weight (N=1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tongue carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel 60/10 Primary (N=117) | Prasugrel 30/7.5 Primary (N=122) | Prasugrel 30/5 Primary (N=133) | Clopidogrel 300/75 Primary (N=135) | Prasugrel 30/5 Low Weight/Elderly (N=91) | Clopidogrel 300/75 Low Weight/Elderly (N=93) | Clopidogrel 300/75 No Weight (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 4 (6) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 8 (8) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enema administration (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days